CLINICAL TRIAL: NCT02089243
Title: Prospective Randomized Controlled Study of Vagus Nerve Stimulation Therapy in the Patients With Medically Refractory Medial Temporal Lobe Epilepsy; Controlled Randomized Vagus Nerve Stimulation Versus Resection (CoRaVNStiR)
Brief Title: Controlled Randomized Vagus Nerve Stimulation (VNS) Therapy Versus Resection (CoRaVNStiR)
Acronym: CoRaVNStiR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xijing-009
Record Dates: First submitted 2013-04-10; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Epilepsy
Keywords: Epilepsy,Temporal Lobe; Brain Diseases
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe; Brain Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vagus nerve stimulation therapy (Experimental): Surgical follow-up typically occurred 2 weeks postoperatively and, subsequently, on a variable schedule as indicated. The adjustments in device parameters were performed, individually, and solely at the discretion of the primary epileptologist with a formal protocol guiding changes. Retrospective chart review was performed to collect follow-up and outcome data. At the time of last available clinical follow-up, the following data were collected: mean weekly seizure frequency (from seizure logs kept by caretakers or patient or caretaker report averaged of the last 3 months prior to ﬁnal follow-up), complications of VNS therapy, duration of VNS therapy, timing and all subsequent surgical procedures.
  Interventions: Procedure: Vagus nerve stimulation therapy
- Resective surgery (Experimental): The type of surgery performed consisted of standard anterior temporal lobectomy, electrocorticography tailored temporal lobectomy, anteromedial temporal lobectomy, transcortical or transsylvian or subtemporal selective amygdalohippocampectomy, temporal lobe disconnection and hippocampal transection.
  Interventions: Procedure: Resective surgery

INTERVENTIONS:
Procedure: Vagus nerve stimulation therapy — The adjustments in device parameters were performed, individually, and solely at the discretion of the primary epileptologist with a formal protocol guiding changes.
  Arms: Vagus nerve stimulation therapy
Procedure: Resective surgery — The experienced neurosurgery are responsible for the selection of surgical techniques employed for medically refractory medial temporal lobe epilepsy that provide an effective treatment with significant preservation of neurological function and acceptable surgical risks.
  Arms: Resective surgery

SUMMARY:
Background: There are a variety of treatment options for medically refractory medial temporal lobe epilepsy. Evidence from randomized trials indicates vagus nerve stimulation therapy can be used as a proven therapy for medically refractory medial temporal lobe epilepsy. Resective surgery is one of the most commonly used methods to treat medically refractory medial temporal lobe epilepsy. The aim of this study is to compare the effects of vagus nerve stimulation therapy and resective surgery in the treatment of the medically refractory medial temporal lobe epilepsy.

Methods/Design: In this article, we report the design and protocol of a randomized controlled trial to treat medically refractory medial temporal lobe epilepsy with vagus nerve stimulation therapy or resective surgery. In total, 40 patients aged 12 to 60 years with medically refractory medial temporal lobe epilepsy will be assessed. There are two treatment groups. These patients are randomly assigned to be in one of the following two treatment groups, i.e. 1) undergo temporal lobe resection group, 2) receive vagus nerve stimulation therapy group. The primary outcome is to assess whether vagus nerve stimulation produces a reduction in mean monthly seizure frequency that is comparable to resection at 3 months, 6 months, 9 months and 12 months of follow-up. The secondary outcomes include the neuropsychological, seizure severity, seizure type, quality of life, mood assessment, operative and postoperative complications and long-term side effects, compared to resection.

Discussion: The result of this trial will assess the efficacy of using vagus nerve stimulation therapy or resective surgery to treat medically refractory medial temporal lobe epilepsy, and to determine a better therapy for treating medically refractory medial temporal lobe epilepsy.

DETAILED DESCRIPTION:
Published data suggest that patients with temporal lobe epilepsy who continue to experience seizures after trials of two or three antiepileptic drugs are unlikely to become seizure-free with further attempts at resection. Such patients may experience poor quality of life and functional outcomes from continuing seizures and the adverse effects associated with further attempts at resection. Vagus nerve stimulation is a minimally invasive treatment for epilepsy with well-established effectiveness as an adjunctive treatment for partial seizures refractory to resection, but there are no vagus nerve stimulation is a minimally invasive treatment for epilepsy with well-established effectiveness as an adjunctive treatment for partial seizures refractory to resection, but there are no controlled randomized clinical trials comparing the effectiveness of Vagus Nerve Stimulation therapy with resection in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Presurgical candidates with pharmacoresistant partial seizures despite optimal medical treatment and history of medically refractory medial temporal lobe epilepsy
* Age above 12 years, below 60 years
* Average of 2 partial seizures per month during a baseline of 2 months
* Recording of seizures must have been done in a prospective manner using standard seizure diaries
* Video-EEG characteristics showing temporal lobe seizure onset (left-sided or right-sided seizure onset) in at least one recorded habitual seizure
* Presence of a structural abnormality in the medial temporal lobe, suggestive of hippocampal sclerosis as evidenced by optimum MRI
* Women of child-bearing age will be required to use a reliable method of contraception during the study duration,
* Patient must be able to provide reliable seizure counts using seizure diaries and to complete the evaluations specified in the study procedures flow chart
* Patient must provide written informed consent, or legal guardian must give written permission and the minor provide written assent.

Exclusion Criteria:

* Extratemporal epilepsy; multifocal epilepsy; evidence of bilateral medial medically refractory medial temporal lobe epilepsy
* MRI evidence of potentially epileptogenic lesions outside the medial temporal lobe such as dysplasias, tumours or cavernomas
* Prior resective intracranial surgery
* Patients who are candidates for invasive video-EEG recording or have previously been investigated with invasive video-EEG recording
* Patients who previously underwent any other type of neurostimulation for treating epilepsy
* Patients who unable to fill in questionnaires and comply with protocol requirements
* Progressive neurological or medical conditions
* Medical or psychiatric conditions precluding surgery or compliance
* Patients taking antidepressant medication
* Pregnancy at study onset
* Previous (within the last 3 months), ongoing or planned participation in other treatment study protocols for epilepsy
* Contraindication for intracranial surgery
* Contraindication for Vagus Nerve Stimulation Therapy
* Patient has had a bilateral or left cervical vagotomy, currently uses, or is expected to use during the study, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy,
* A VNS Therapy System implant would (in the investigator's judgment) pose an unacceptable surgical or medical risk for the patient
* Patient is expected to require full body magnetic resonance imaging during the clinical study
* Patient has had a previous VNS Therapy System implant.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
seizure frequency | 3 months

SECONDARY OUTCOMES:
neuropsychological examination | 12 months
responder rates | during 3 month intervals
mean seizure free interval | during 3 month intervals
seizure severity | during 3-month intervals
quality of life | 3 months, 6 months, 9 months and 12 months
complications | during twelve months after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Yanchun YC Deng, MD, PhD, Study Director — the Department of Neurology, Xijing Hospital
Locations (1):
- the Department of Neurology, Xijing Hospital, Xi'an, Shaanxi, China